CLINICAL TRIAL: NCT05755074
Title: Ablation of Typical Right Atrial Flutter Through the Arm: Evaluation of Safety, Feasibility, and Efficacy
Brief Title: Ablation of Typical Right Atrial Flutter
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hartford Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HHC20200300
Record Dates: First submitted 2020-10-20; First posted 2023-03-06 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Atrial Flutter
Keywords: ablation; safety; efficacy
MeSH Terms: conditions — Atrial Flutter

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ablation through upper extremity (Experimental): Ablation through arm
  Interventions: Procedure: Ablation through left arm
- Ablation through femoral vein (Active Comparator): Ablation through vein
  Interventions: Procedure: Ablation through femoral vein

INTERVENTIONS:
Procedure: Ablation through left arm — Ablation through left arm
  Arms: Ablation through upper extremity
Procedure: Ablation through femoral vein — Ablation through femoral vein
  Arms: Ablation through femoral vein

SUMMARY:
Typical atrial flutter ablation involving forming a line of block across the cavotricuspid isthmus in the right atrium has become a commonly performed procedure and is considered a class I indicated procedure for patients who wish to pursue maintenance of sinus rhythm. The ablation generally involves 2-3 catheters and is typically performed through the femoral vein(s). After the ablation procedure, the patient is placed on bed rest for 4 hours, and typically discharged home the same day on oral anticoagulation.

Catheter technology has improved over the past several years allowing for more rapid ablation with shorter procedure times. Ultrasound has also become more routinely used when obtaining venous access for the patient.

To date, ablation of typical atrial flutter through the left or right arm has not been reported. Diagnostic electrophysiology studies have been performed through the arm and AV node ablation has also been reported from the cephalic, internal jugular, axillary and subclavian veins. The potential benefits include shorter recovery time, reduced risk of retroperitoneal bleed, and the avoidance of access complications from the groin.

This study aims to evaluate the safety, feasibility, and efficacy of performing typical atrial flutter ablation through the arm.

Specifically, the study will aim to:

1. Compare the recovery time immediately after the procedure using upper extremity access compared to the standard approach.
2. Compare the success rate of patients that undergo ablation of typical atrial flutter through the upper extremity venous system (experimental approach) to the standard approach (i.e., through the femoral vein(s). Success will be defined as ablation that leads to evidence for bidirectional block across the right atrial cavotricuspid isthmus.
3. Establish what the potential complications are from performing typical atrial flutter through the left or right arm. The left arm will be the preferred site for access because of less tortuosity to reach the heart. If one side cannot be accessed the alternate arm will be used, but will be left to the discretion of the operator. The operator will have the discretion to switch to a femoral approach at any time.
4. Compare the complication rates of the experimental approach evaluated by the inability to access the vein, and other complications (e.g., bleeding, vein thrombosis, heart perforation) from accessing the vein in the arm to the complication rates of the standard approach.
5. Compare long term (i.e., 1 month and 1 year) success of the experimental approach vs. the standard approach as assessed by maintenance of normal sinus rhythm, without recurrent typical right atrial flutter with in person visits and phone call or chart evaluations.
6. Compare pain severity of the insertion site between the experimental and standard approaches.

ELIGIBILITY:
Inclusion Criteria:

* Referred to the EP lab for typical right atrial flutter ablation as an outpatient
* Bodyweight of 50Kg (110 lb) or above
* Documented typical atrial flutter by 12 lead EKG or telemetry

Exclusion Criteria:

* Bodyweight less than 50 Kg
* Inability to provide consent
* Presence of pacemaker or defibrillator with transvenous leads
* Inpatient admission

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-10-28 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Recovery time | Immediately after procedure
  Recovery time after procedure is defined as clock time when the patient is deemed ready for discharge minus clock time when the patient's procedure has ended

SECONDARY OUTCOMES:
Success rate | Measured during procedure
  Percentage of patients with ablation leading to evidence of bidirectional block
Frequency of complications | Measured during procedure
  Frequency of complications that arise from performing ablation for atrial flutter through the left or right arm.
Complication rate | Measured during procedure
  Percentage of patient with complications after ablation for atrial flutter
One month success rate | Measured at one month after ablation
  Percentage of patients maintaining normal sinus rhythm, without recurrent typical right atrial flutter
One year success rate | Measured at one year after ablation
  Percentage of patients maintaining normal sinus rhythm, without recurrent typical right atrial flutter
Pain severity scale | Measured once at discharge
  The pain severity scale measures pain on a scale of 1 to 10 (10 being extremely painful, 1 being no pain). Patients will be asked "how much pain are you feeling at the site in which the catheter was inserted?" and will give an answer from 0 to 10, as described above.

CONTACTS AND LOCATIONS:
Overall Officials: Aneesh Tolat, MD, Principal Investigator — Hartford Hospital
Locations (1):
- Hartford Hospital, Hartford, Connecticut, United States